CLINICAL TRIAL: NCT06213077
Title: To Determine the Potentiating Effects of Berkeley Life Foundation Nitric Oxide Capsules in Supporting Healthy Sexual Function in Men on an Existing Treatment Plan But Who Are Experiencing Occasional Unsatisfactory Erections.
Brief Title: The Effects of a Nitrate Supplementation on Erectile Function
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: RHA Investments Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: #EDSupp23
Record Dates: First submitted 2023-12-29; First posted 2024-01-19 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Erectile Dysfunction
Keywords: Erectile Dysfunction; Nitric Oxide
MeSH Terms: conditions — Erectile Dysfunction | interventions — Nitric Oxide; Tadalafil

STUDY DESIGN:
Intervention Model Description: IRB approved, double blind placebo-controlled crossover study
Who Masked: Participant, Investigator
Masking Description: IRB approved, double blind placebo-controlled crossover study. Control product (Tadalafil) open label. Nitric Oxide and placebo products labelled Sample 1 and Sample 2.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nitric Oxide (Active Comparator): Upon enrollment, patients will complete the IIEF questionnaire, EHS Score questionnaire and the Quality of Life survey.
  Patients will be sent home with instructions to take 2 Berkeley Life capsules once daily (in this case Active NO), in combination with their existing treatment protocol (Tadalafil) and then return on day 60, returning all unused test product.
  After 60 days of taking the active ingredient + tadalafil, patients will repeat the IIEF questionnaire, EHS Score questionnaire and the Quality of Life survey.
  After a 4 week wash out, patients will be crossed over to the placebo group and given the other combination.
  After 60 days of both combinations, placebo and active, patients will repeat the IIEF questionnaire, EHS Score questionnaire and the Quality of Life survey
  Interventions: Dietary Supplement: Nitric Oxide; Drug: Tadalafil
- Placebo (Placebo Comparator): Upon enrollment, patients will complete the IIEF questionnaire, EHS Score questionnaire and the Quality of Life survey.
  Patients will be sent home with instructions to take 2 Berkeley Life capsules once daily (in this case the placebo), in combination with their existing treatment protocol (Tadalafil) and then return on day 60, returning all unused test product.
  After 60 days of taking the placebo + tadalafil, patients will repeat the IIEF questionnaire, EHS Score questionnaire and the Quality of Life survey.
  After a 4 week wash out, patients will be crossed over to the active group and given the other combination.
  After 60 days of each combination, placebo and active, patients will repeat the IIEF questionnaire, EHS Score questionnaire and the Quality of Life survey
  Interventions: Drug: Tadalafil; Other: Placebo

INTERVENTIONS:
Dietary Supplement: Nitric Oxide — Naturally produced and found in many different kinds of cells and organ systems, NO is an integral molecule in regulating blood pressure and maintaining a healthy cardiovascular system. NO produced or generated in the vasculature then diffuses into the underlying smooth muscle causing these muscles to relax. This results in vasodilation, causing a reduction in systemic blood pressure and an increase in blood flow and oxygen delivery to specific vascular beds.
  Other Names: Berkeley Life
  Arms: Nitric Oxide
Drug: Tadalafil — Vasodilator which treats erectile dysfunction and enlarged prostate (benign prostatic hyperplasia). It can also treat high blood pressure in the lungs (pulmonary arterial hypertension).
Other: Placebo — Nitric Oxide Placebo Compound
  Arms: Placebo

SUMMARY:
Twenty (20) individuals to be recruited from Ballantyne Medical Associates in Charlotte, NC, without any significant chronic medical history. These patients are general patients for primary care that meet inclusion criteria. Patients will be screened and enrolled by Dr. Bauer and his delegated research staff upon patient consult. Patients will be informed of the purpose of the study including risks, benefits, and alternative treatments to the study. After the potential participants have been given the opportunity to ask questions and have their questions answered, they will be asked to sign an informed consent prior to any study-specific procedures being performed.

Blinded test product will be randomly assigned to study subjects. Test group 1 will be dosed with a placebo capsule taken two capsules once daily Test group 2 will be dosed with Berkeley Life capsules taken two capsules once daily. At baseline, prior to crossover to the other treatment, and at the study's conclusion, NO levels will be monitored using salivary nitric oxide test strips. Both test groups will remain on their existing treatment protocol throughout the study.

DETAILED DESCRIPTION:
Patients will be consented and enrolled in the study. A complete medical history and focused physical examination will be conducted and documented and NO levels will be measured using salivary test strips.

Twenty (20) patients with low NO levels will be enrolled and will be randomly assigned to group 1 or group 2.

Once enrolled, patients will be required to complete a subjective questionnaire (the International Index of Erectile Function (IIEF)), EHS Score questionnaire and a Quality of Life (QOL) survey. Patients will be instructed to take 2 Berkeley Life capsules once daily or the placebo based on randomization. The (IIEF) was developed by Rosen and colleagues in 1997 as a multidimensional, 15-item, self-administered questionnaire with the goal of assessing five domains of male sexual function including erectile function, orgasmic function, sexual desire, intercourse satisfaction, and overall satisfaction. The erectile function domain of the IIEF (IIEF-EF) contains 6 questions which the patient answers on a scale from 1 (never or almost never) to 5 (almost always or always), providing a total score of 6 to 30 points. The questions concern erectile frequency, firmness, penetration ability, maintenance frequency, maintenance ability, and erection confidence. Based on a controlled study of 1,151 men taking sildenafil in order to establish cutoff scores for the IIEF-EF, a score of 26 or greater is defined as normal function, mild ED is a score from 22 to 25, mild to moderate ED 17 to 21, moderate ED 11 to 16, and severe ED 6 to 10.

Patients will be sent home with instructions to take 2 Berkeley Life capsules once daily in combination with their existing treatment protocol and then return on day 60, returning all unused test product.

The subject should be willing to self-administer 2 capsules daily and be willing to, upon waking in the AM, self-test with strip and record on a pre-print sheet the test strip color, followed by self-administration of capsule(s) and then at 2 hours self-test again and record on a pre-print sheet the test strip color.

Upon the return visit, patients will be crossed over after a 4 week wash out and given the other test group combination.

After 60 days of each combination, placebo and active, patients will repeat the IIEF questionnaire, EHS Score questionnaire and the Quality of Life survey.

The remaining product will be collected, and patients released from the study. Data will be collected on Case Report Forms.

ELIGIBILITY:
Inclusion Criteria:

* Subjects Male between the ages of 40 and 65
* Subjects looking to support healthy sexual function who have been undergoing treatment to support healthy erections for at least 90 days with unsatisfactory results and whose nitric oxide levels are suboptimal based on an easy-to-use, self-check saliva strip that provides immediate, real-time, actionable feedback.
* Patients who are able to sign informed consent.

Exclusion Criteria:

* Patients who are not considered medically stable (history of drug or alcohol dependency or having experienced health issues which could prevent experiencing a healthy erection).
* Patients with any known allergy to ingredients of capsule.
* Patients currently taking organic nitrates for acute angina
* Patients who do not or cannot tolerate PDE5 inhibitors
* Patients are unwilling or unable to provide informed consent.

Ages: 40 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 20 (Estimated)
Dates: Start 2023-12-12 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-05-30 (Estimated)

PRIMARY OUTCOMES:
International Index of Erectile Function | Initial, 2 months post first arm, 2 months post second arm
  The (IIEF) was developed by Rosen and colleagues in 1997 as a multidimensional, 15-item, self-administered questionnaire with the goal of assessing five domains of male sexual function including erectile function, orgasmic function, sexual desire, intercourse satisfaction, and overall satisfaction [17]. The erectile function domain of the IIEF (IIEF-EF) contains 6 questions which the patient answers on a scale from 1 (never or almost never) to 5 (almost always or always), providing a total score of 6 to 30 points. The questions concern erectile frequency, firmness, penetration ability, maintenance frequency, maintenance ability, and erection confidence. Based on a controlled study of 1,151 men taking sildenafil in order to establish cutoff scores for the IIEF-EF, a score of 26 or greater is defined as normal function, mild ED is a score from 22 to 25, mild to moderate ED 17 to 21, moderate ED 11 to 16, and severe ED 6 to 10.
Erection Hardness Score | Initial, 2 months post first arm, 2 months post second arm
  The Erection Hardness Scale (EHS) involves a 1-4 response to a single question to assess firmness of erection, where 3 is sufficient for penetration and 4 is a rigid erection

SECONDARY OUTCOMES:
SF-36 Quality of Life Questionnaire | Initial, 2 months post first arm, 2 months post second arm
  The 36-Item Short Form Health Survey (SF-36) in 1992. SF-36 is a set of generic, coherent, and easily administered quality-of-life measures. These measures rely upon patient self-reporting and have been widely used.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Bauer, Principal Investigator — Onsite Clinical Solutions
Locations (1):
- OnSite Clinical Solutions, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No